CLINICAL TRIAL: NCT07058077
Title: An Operationally Seamless Phase 2/3 Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Enlicitide Decanoate in Pediatric Participants With Heterozygous Familial Hypercholesterolemia
Brief Title: A Study of Enlicitide Decanoate (MK-0616, an Oral PCSK9 Inhibitor) in Children and Adolescents With Heterozygous Familial Hypercholesterolemia (MK-0616-029)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0616-029; U1111-1314-5796 (Registry Identifier: UTN); 2024-519068-42-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Heterozygous Familial Hypercholesterolemia (HeFH)
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Intervention Model Description: There are two parts of the study. Part A is a non randomized single treatment group. Part B is randomized parallel treatment groups. Participants who complete either part are then eligible to enroll in an open label extension (single group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A and the extension period are open-label. Part B is double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Enlicitide Decanoate (Experimental): Participants receive enlicitide decanoate orally once daily (QD) at a dosage determined by age for up to 2 weeks.
  Interventions: Drug: Enlicitide Decanoate
- Part B: Enlicitide Decanoate (Experimental): Participants receive enlicitide decanoate QD at a dosage determined by age for up to 24 weeks.
  Interventions: Drug: Enlicitide Decanoate
- Part B: Placebo (Placebo Comparator): Participants receive placebo orally QD for up to 24 weeks.
  Interventions: Drug: Placebo
- Open-Label Extension: Enlicitide Decanoate (Experimental): Participants who complete either Part A or Part B may enroll in this open-label extension arm. Participants in the extension arm receive enlicitide decanoate QD at a dosage determined by age for up to 3 years.
  Interventions: Drug: Enlicitide Decanoate

INTERVENTIONS:
Drug: Enlicitide Decanoate — Enlicitide decanoate taken by mouth
  Other Names: MK-0616; Enlicitide
  Arms: Open-Label Extension: Enlicitide Decanoate; Part A: Enlicitide Decanoate; Part B: Enlicitide Decanoate
Drug: Placebo — Placebo tablet matched to enlicitide decanoate taken by mouth
  Arms: Part B: Placebo

SUMMARY:
This study is designed to learn if enlicitide decanoate is safe and effective to treat children and adolescents with heterozygous familial hypercholesterolemia (HeFH) and high amounts of low-density lipoprotein cholesterol (LDL-C) in the blood.

The goals of this study are to learn about the safety of enlicitide and if children tolerate it, what happens to enlicitide in a child's body over time, and if enlicitide works to lower cholesterol levels in children more than a placebo.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to:

* Has possible or definite diagnosis of HeFH based on a locally accepted diagnostic algorithm or diagnosis by genetic testing results
* Has a fasted LDL-C value (evaluated by the central laboratory) that is ≥130 mg/dL
* Is receiving either an optimized daily dose of statin (± nonstatin LLT); or a nonstatin LLT with documented intolerance to at least 2 different statins or refusal of statin therapy by the participant or legally acceptable representative
* Is on a stable dose of all background LLTs for at least 30 days prior to screening, with no medication or dose changes planned during participation in Part A or Part B

Exclusion Criteria:

Exclusion criteria include, but are not limited to:

* Has a history of homozygous FH based on genetic or clinical criteria, or history of known compound heterozygous FH, or double heterozygous FH
* Has a history of nephrotic syndrome
* Has any clinically significant malabsorption condition based on principal investigator assessment
* Was previously treated/is being treated with certain other cholesterol lowering medications, including proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors without adequate washout

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2033-12-04 (Estimated); Study Completion 2037-01-23 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximum Plasma Concentration (Cmax) of Enlicitide | At designated timepoints (up to 24 hours postdose on day 14)
  Blood samples will be collected to determine the Cmax of enlicitide.
Part A: Area Under the Concentration-Time Curve from 0 to 24 Hours (AUC0-24) of Enlicitide | At designated timepoints (up to 24 hours postdose on day 14)
  Blood samples will be collected to determine the AUC0-24 of enlicitide.
Part B: Percent Change from Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline and Week 24
  Blood samples will be collected to determine the percent change from baseline in LDL-C.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 188 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 180 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Part B: Percent Change from Baseline in Apolipoprotein B (ApoB) | Baseline and week 24
  Blood samples will be collected to determine the percent change from baseline in apolipoprotein B.
Part B: Percent Change from Baseline in Non-High-Density Lipoprotein Cholesterol (non-HDL-C) | Baseline and week 24
  Blood samples will be collected to determine the percent change from baseline in non-HDL-C.
Part B: Percent Change from Baseline in Lipoprotein (a) (Lp(a)) | Baseline and week 24
  Blood samples will be collected to determine the percent change from baseline in Lp(a).
Part B: Percentage of Participants With LDL-C <130 mg/dL at Week 24 | Week 24
  The percentage of participants with LDL-C <130 mg/dL at week 24 will be reported.
Part B: Percentage of Participants With ≥50% LDL-C LDL-C Reduction from Baseline at Week 24 | Baseline and week 24
  The percentage of participants with ≥50% LDL-C reduction from baseline at week 24 will be reported.
Part B: Percentage of Participants With LDL-C <100 mg/dL at Week 24 | Week 24
  The percentage of participants with LDL-C <100 mg/dL at week 24 will be reported.
Change in Carotid Intima-media Thickness (cIMT) | Baseline and week 24
  Ultrasound measurements will be performed to determine the change from baseline in cIMT.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- United States (4):
  - Nemours/Alfred I. duPont Hospital for Children ( Site 0001), Wilmington, Delaware
  - Children's National Medical Center ( Site 0015), Washington D.C., District of Columbia
  - Excel Medical Clinical Trials ( Site 0008), Boca Raton, Florida
  - Children's Healthcare of Atlanta Cardiology ( Site 0026), Atlanta, Georgia
- Brazil (2):
  - Universidade Federal Do Ceara ( Site 0201), Fortaleza, Ceará
  - Incor - Instituto do Coracao ( Site 0200), São Paulo
- China (2):
  - Beijing Anzhen Hospital. Capital Medical University ( Site 1917), Beijing, Beijing Municipality
  - The Children's Hospital of Zhejiang University School of Medicine ( Site 1905), Hangzhou, Zhejiang
- Colombia (4):
  - Clinica de la Costa S.A.S. ( Site 0400), Barranquilla, Atlántico
  - Oncomédica S.A.S ( Site 0401), Montería, Departamento de Córdoba
  - Fundación Cardiovascular de Colombia ( Site 0402), Piedecuesta, Santander Department
  - Fundacion Valle del Lili ( Site 0403), Cali, Valle del Cauca Department
- New Zealand Clinical Research (Christchurch) ( Site 1700), Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com